CLINICAL TRIAL: NCT03356951
Title: Analysis of Patients Who Underwent Ankle Replacement and Simultaneous Subtalar Fusion by Biomechanical and Clinical Evaluation
Brief Title: Gait Analysis Following Total Ankle Replacement and Subtalar Fusion
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: MAT
Record Dates: First submitted 2017-11-19; First posted 2017-11-29 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Ankle Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lateral approach group: TAR through lateral approach and subtalar fusion
  Interventions: Procedure: TAR through lateral approach and subtalar fusion
- Anterior approach group: TAR through anterior approach and subtalar fusion
  Interventions: Procedure: TAR through anterior approach and subtalar fusion

INTERVENTIONS:
Procedure: TAR through anterior approach and subtalar fusion — Simultaneous total ankle replacement through anterior approach and subtalar fusion
  Other Names: Hintegra ankle system
  Groups: Anterior approach group
Procedure: TAR through lateral approach and subtalar fusion — Simultaneous total ankle replacement through lateral approach and subtalar fusion
  Other Names: Zimmer TM (Trabecular Metal ) Total Ankle
  Groups: Lateral approach group

SUMMARY:
Subtalar fusion is commonly performed in post-traumatic subtalar osteoarthritis, rheumatoid arthritis, posterior tibial tendon dysfunction, tarsal coalition and primary subtalar osteoarthritis. Patients with osteoarthritis or severe dysfunction involving both the ankle and the subtalar joint may benefit from an tibiotalocalcaneal fusion (TTC) or an ankle replacement and subtalar fusion. With the development of new prosthetic designs and of surgical techniques, total ankle replacements (TAR) became a reasonable alternative to fusion with functional and quality of life improvements. A gait analysis of patients that underwent TAR and simultaneous subtalar fusion allows to study with precision and reliability the ankle range of motion (ROM). On the contrary, in healthy subjects or in patients that underwent isolated TAR this is not possible because the ankle ROM is influenced by the ROM of the subtalar joint in such a way that it is not possible to analyze the two joints separately. Also, excluding the role of the subtalar joint, it is possible to accurately analyze and compare the consequences on ankle kinematics of two different prosthetic designs.

DETAILED DESCRIPTION:
Patients who previously have underwent TAR and simultaneous subtalar fusion are retrospectively reviewed. Minimum follow-up after the surgery is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent ankle prosthesis (Hintegra ankle system, Zimmer Trabecular Metal Total Ankle) and simultaneous fusion of the subtalar joint with at least 12 months of follow-up willing and capable of adhering to postoperative clinical protocols and functional evaluations and who have signed a specific informed consent form approved by the Ethics Committee
* Males or females aged between 20 and 80 years old.
* Patients with diagnosis of primary not-inflammatory degenerative articular disease

Exclusion Criteria:

* Patients with Body Mass Index (BMI)> 35.
* Patients with active or suspected latent periprosthetic infection
* Patients who underwent revision surgery.
* Prosthesis of the hip, knee or ankle, homolateral or contralateral.
* Fusion failure of subtalar joint.
* Patients with chronic heart failure (NYHA stage> 2)
* Presence of neurological disorders, neuromuscular disorders or other major musculoskeletal pathologies
* Cognitive deficits.
* Impossibility to match questionnaires due to cognitive disorders or language dysfunctional disorders

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent simoultanous total ankle replacement and subtalar fusion
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Gait analysis | 1 day
  Differences in functional scores obtained by Mini-lab stereophotogrammetry-based Gait Analysis for Lower Limbs

SECONDARY OUTCOMES:
VAS (Visual Analog Scale) | 1 day
  Differences in Pain Scores on the Visual Analog Scale
AOFAS | 1 day
  Differences in Functional Scores on the American Orthopaedic Foot and Ankle Society Score
Short Form Health Survey (SF-12) | 1 day
  Differences in Health Scores on the 12-Item Short Form Health Survey

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy

REFERENCES:
- [Derived] Usuelli FG, Indino C, Leardini A, Manzi L, Ortolani M, Caravaggi P. Range of motion of foot joints following total ankle replacement and subtalar fusion. Foot Ankle Surg. 2021 Feb;27(2):150-155. doi: 10.1016/j.fas.2020.03.015. Epub 2020 Apr 27. PMID 32381452